CLINICAL TRIAL: NCT01214109
Title: A Multiple Dose Bioequivalence Study of Pramipexole With Increasing Doses (0.375mg to 1.5mg q.d.) of Oral Extended Release (ER) Tablet in Two-way Cross-over Comparison of 0.375mg Extended Release Tablet q.d. Versus 0.125mg Immediate Release (IR) Tablet t.i.d and 1.5 mg Extended Release Tablet q.d. Versus 0.5mg Immediate Release Tablet t.i.d. in Chinese Healthy Male Volunteers
Brief Title: Multiple Dose Bioequivalence Study of Pramipexole Extended Release in Chinese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 248.665
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
MeSH Terms: interventions — Pramipexole

ARMS (2):
- pramipexole extended release (Experimental): 0.375mg once per day for 5 days (cross-over), 0.75mg once per day for 5 days (up-titration), 1.5mg once per day for 5 days (cross-over)
  Interventions: Drug: pramipexole extended release; Drug: pramipexole immediate release
- pramipexole immediate release (Active Comparator): 0.125mg three times a day for 5 days (crossover), 0.5mg three times a day for 5 days (cross over)
  Interventions: Drug: pramipexole extended release; Drug: pramipexole immediate release

INTERVENTIONS:
Drug: pramipexole extended release — 0.375mg once per day for 5 days (cross-over), 0.75mg once per day for 5 days (up-titration), 1.5mg once per day for 5 days (cross-over)
  Arms: pramipexole immediate release
Drug: pramipexole extended release — 0.375mg once per day for 5 days (cross-over), 0.75mg once per day for 5 days (up-titration), 1.5mg once per day for 5 days (cross-over)
  Arms: pramipexole extended release
Drug: pramipexole immediate release — 0.125mg three times a day for 5 days (crossover), 0.5mg three times a day for 5 days (cross over)
  Arms: pramipexole immediate release
Drug: pramipexole immediate release — 0.125mg three times a day for 5 days (crossover), 0.5mg three times a day for 5 days (cross over)
  Arms: pramipexole extended release

SUMMARY:
To establish bioequivalence at steady state of:

1)0.375 mg pramipexole extended release tablet q.d. in fasted status versus 0.125 mg pramipexole Immediate release tablet t.i.d. in fasted status 2)1.5 mg pramipexole extended release tablet q.d. in fasted status versus 0.5 mg pramipexole Immediate release tablet t.i.d. in fasted status

To investigate dose proportionality of pharmacokinetics parameters for:

1)pramipexole extended release dosage of 0.375 to 1.5 mg q.d.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, clinical laboratory tests
2. Age older than or equal 18 and Age younger than or equal 40 years
3. Body Mass Index larger than or equal 19 and Body Mass Index less than or equal 24kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including Pulse Rate and electrocardiogram) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (longer than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial up to 7 days before the start of drug administration in the study or during the study period
11. Participation in another trial with an investigational drug within one months prior to administration or during the trial
12. Smoker (more than 10 cigarettes or more than 3 cigars or more than 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 40 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Any positive results in hepatitis B surface antigen (HBsAg), anti hepatitis B core (HBc) antibodies, anti hepatitis C virus (HCV) antibodies and human immunodeficiency virus (HIV) test

    Exclusion criteria specific for this study:
20. Hypersensitivity to pramipexole or other dopamine agonists
21. Supine blood pressure at screening of systolic<100 mmHg and diastolic < 60 mmHg, or symptomatic orthostatic hypotension (i. .e. clinical symptoms of orthostatic hypotension associated with a decline >=20 mmHg in systolic BP and a decline >=10 mmHg in diastolic BP, at one minute after standing compared to the previous supine systolic and diastolic BP obtained after 5 minutes of quiet rest)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 248.665.86002 Boehringer Ingelheim Investigational Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 subjects were equally randomised to one of two groups / sequences, and in general terms, ABCD or BADC. Hence, 12 subjects were in group ABCD and 12 in BADC. All 24 subjects received all treatments, A, B, C, D. The numbers presented in the milestone are by overall treatment, A, B, C or D.
Groups:
- 0.375 mg q.d.Extended Release (ER): 0.375mg once daily (q.d.) of oral extended release (ER) tablet of pramipexole
- 0.125 mg t.i.d. Immediate Release (IR): 0.125mg thrice daily (t.i.d) of immediate release (IR) tablet of pramipexole
- 1.5 mg q.d. ER: 1.5mg once daily (q.d.) of oral extended release (ER) tablet of pramipexole
- 0.5 mg t.i.d. IR: 0.5mg thrice daily (t.i.d) of immediate release (IR) tablet of pramipexole
Period: Overall Study
Arm/Group | 0.375 mg q.d.Extended Release (ER) | 0.125 mg t.i.d. Immediate Release (IR) | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Started | 24 | 24 | 24 | 24
Completed | 24 | 24 | 24 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: 24 subjects were equally randomised to one of two groups / sequences, and in general terms, ABCD or BADC. Hence, 12 subjects were in group ABCD and 12 in BADC. All 24 subjects received all treatments, A, B, C, D. The numbers presented are by overall treatment.
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Pramipexole in Plasma at Steady State Over 24 Hours (AUC0-24,ss); in Case of ER up to the Time Point of Next Dosing (AUCtau,ss) for Pharmacokinetic (PK) Population (All Subjects)
Description: AUC0-24,ss = area under the plasma concentration-time curve between 0 and 24 hours at steady state. AUCtau,ss = area under the plasma concentration-time curve over a dosing interval at steady state
Time Frame: 27 days
Population: PK population - Subjects with values for AUC0-24,ss for IR and values for AUCtau,ss for ER
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 0.375 mg q.d.ER: 0.375mg once daily (q.d.) of oral extended release (ER) tablet of pramipexole
- 0.125 mg t.i.d. IR: 0.125mg thrice daily (t.i.d) of immediate release (IR) tablet of pramipexole
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 23 | 24
ng*h/mL | 6.20 (29.7) | 7.50 (21.5) | 19.1 (113) | 20.4 (104)
Statistical Analysis 1: Comparison: 0.375 mg q.d.ER vs 0.125 mg t.i.d. IR; 0.125 mg t.i.d. IR is the reference treatment, 0.375 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 82.62, 90% CI [74.45 to 91.69]
Statistical Analysis 2: Comparison: 1.5 mg q.d. ER vs 0.5 mg t.i.d. IR; 0.5 mg t.i.d. IR is the reference treatment, 1.5 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 96.17, 90% CI [69.33 to 133.42]

2. Primary Outcome: Area Under the Concentration-time Curve of Pramipexole in Plasma at Steady State Over 24 Hours (AUC0-24,ss); in Case of ER up to the Time Point of Next Dosing (AUCtau,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: as for outcome 1
Time Frame: 27 days
Population: PK population excluding subjects with reported emesis - Subjects with values for AUC0-24,ss for IR and values for AUCtau,ss for ER, excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
ng*h/mL | 6.64 (19.6) | 7.44 (22.6) | 24.8 (34.6) | 27.4 (40.4)
Statistical Analysis 1: Comparison: 0.375 mg q.d.ER vs 0.125 mg t.i.d. IR; 0.125 mg t.i.d. IR vs. 0.375 mg q.d. ER 0.125 mg t.i.d. IR is the reference treatment, 0.375 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 88.01, 90% CI [80.76 to 95.92]
Statistical Analysis 2: Comparison: 1.5 mg q.d. ER vs 0.5 mg t.i.d. IR; 0.5 mg t.i.d. IR vs. 1.5 mg q.d. ER 0.5 mg t.i.d. IR is the reference treatment, 1.5 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 89.37, 90% CI [81.16 to 98.42]

3. Primary Outcome: Maximum Steady State Concentration (Cmax,ss) for PK Population (All Subjects)
Description: Cmax = maximum observed concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK population - Subjects with values for Cmax,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 24 | 24
ng/mL | 0.416 (25.3) | 0.469 (22.1) | 1.10 (130) | 1.20 (112)
Statistical Analysis 1: Comparison: 0.375 mg q.d.ER vs 0.125 mg t.i.d. IR; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 88.82, 90% CI [79.89 to 98.76]
Statistical Analysis 2: Comparison: 1.5 mg q.d. ER vs 0.5 mg t.i.d. IR; 0.5 mg t.i.d. IR vs. 1.5 mg q.d. ER 0.5 mg t.i.d. IR is the reference treatment, 1.5 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 91.97, 90% CI [60.07 to 140.25]

4. Primary Outcome: Maximum Steady State Concentration (Cmax,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: Cmax,ss = maximum observed concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK population excluding subjects with reported emesis - Subjects with values for Cmax,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
ng/mL | 0.436 (20.6) | 0.463 (22.8) | 1.56 (26.5) | 1.61 (42.6)
Statistical Analysis 1: Comparison: 0.375 mg q.d.ER vs 0.125 mg t.i.d. IR; 0.125 mg t.i.d. IR is the reference treatment, 0.375 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 92.84, 90% CI [83.8 to 102.86]
Statistical Analysis 2: Comparison: 1.5 mg q.d. ER vs 0.5 mg t.i.d. IR; 0.5 mg t.i.d. IR is the reference treatment, 1.5 mg q.d. ER is the test treatment; Test type: Superiority or Other; ANOVA; Ratio of geometric least squares means = 95.05, 90% CI [84.88 to 106.43]

5. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of the Analyte in Plasma (Tmax) for PK Population (All Subjects)
Description: tmax = time of maximum observed plasma concentration
Time Frame: 27 days
Population: PK population - Subjects with values for tmax
Measure: Median (Full Range); unit: hours
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 24 | 24
hours | 4.00 [0.0 to 8.0] | 1.00 [0.500 to 2.00] | 4.00 [0.00 to 8.00] | 1.00 [0.00 to 2.50]

6. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of the Analyte in Plasma (Tmax) for PK Population (Excluding Subjects Due to Emesis)
Description: tmax = time of maximum observed plasma concentration
Time Frame: 27 days
Population: PK population excluding subjects with reported emesis - Subjects with values for t_max excluding subjects with reported emesis
Measure: Median (Full Range); unit: hours
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
hours | 4.00 [1.00 to 8.00] | 1.00 [0.500 to 2.00] | 4.00 [2.00 to 8.00] | 1.00 [0.500 to 2.00]

7. Secondary Outcome: Peak-to-trough Fluctuation (PTF) for PK Population (All Subjects)
Description: PTF = Peak-to-trough fluctuation is measured as a percent
Time Frame: 27 days
Population: PK population - Subjects with values for PTF
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 23 | 24
percent | 112 (29.4) | 86.6 (27.5) | 101 (33.8) | 78.2 (34.5)

8. Secondary Outcome: Peak-to-trough Fluctuation (PTF) for PK Population (Excluding Subjects Due to Emesis)
Description: PTF = Peak-to-trough fluctuation is measured as a percent
Time Frame: 27 days
Population: PK population excluding subjects with reported emesis - Subjects with values for PTF excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
percent | 109 (28.9) | 86.2 (29.1) | 103 (28.3) | 82.5 (24.8)

9. Secondary Outcome: Predose Steady State Concentration of the Analyte Immediately Before Administration of the Next Drug Administration (Cpre,ss) for PK Population (All Subjects)
Description: Cpre,ss = pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose
Time Frame: 27 days
Population: PK population - Subjects with values for Cpre,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 24 | 24
ng/mL | NA (NA) — Not calculated | NA (NA) — Not calculated | NA (NA) — Not calculated | 0.507 (90.4)

10. Secondary Outcome: Predose Steady State Concentration of the Analyte Immediately Before Administration of the Next Drug Administration (Cpre,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: as for outcome 9
Time Frame: 27 days
Population: PK population excluding subjects with reported emesis - Subjects with values for Cpre,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 20 | 21 | 18 | 18
ng/mL | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | 0.487 (105) | 0.616 (57.2)

11. Secondary Outcome: Average Concentration in Plasma Under Steady-state Conditions (Cavg) for PK Population (All Subjects)
Description: Cavg = Average concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK Population - Subjects with values for Cavg
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 23 | 24
ng/mL | 0.259 (29.7) | 0.312 (21.5) | 0.796 (113) | 0.848 (104)

12. Secondary Outcome: Average Concentration in Plasma Under Steady-state Conditions (Cavg) for PK Population (Excluding Subjects Due to Emesis)
Description: Cavg = Average concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK Population excluding subjects with reported emesis - Subjects with values for Cavg excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
ng/mL | 0.277 (19.6) | 0.310 (22.6) | 1.04 (34.6) | 1.14 (40.4)

13. Secondary Outcome: Terminal Half-life of the Analyte in Plasma at Steady State (t1/2,ss) for PK Population (All Subjects)
Description: t1/2,ss - Apparent plasma terminal elimination half-life at steady state
Time Frame: 27 days
Population: PK Population - Subjects with values for t1/2,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 23 | 19 | 24
h | 13.3 (40.7) | 7.69 (28.6) | 14.4 (42.8) | 8.43 (25.3)

14. Secondary Outcome: Terminal Half-life of the Analyte in Plasma at Steady State (t1/2,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: t1/2,ss - Apparent plasma terminal elimination half-life at steady state
Time Frame: 27 days
Population: PK Population excluding subjects with reported emesis - Subjects with values for t1/2,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 19 | 20 | 14 | 18
h | 13.4 (42.6) | 7.68 (30.5) | 14.5 (46.9) | 7.92 (16.6)

15. Secondary Outcome: Minimum Steady State Concentration (Cmin,ss) for PK Population (All Subjects)
Description: Cmin,ss = Minimum observed concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK Population - Subjects with values for Cmin,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 23 | 24
ng/mL | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | 0.478 (95.3)

16. Secondary Outcome: Minimum Steady State Concentration (Cmin,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: Cmin,ss = Minimum observed concentration of the analyte in plasma at steady state
Time Frame: 27 days
Population: PK Population excluding subjects with reported emesis - Subjects with values for Cmin,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
ng/mL | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | NA (NA) — Pharmacokinetic parameters which could not be determined were identified by "not calculated (NC)". | 0.403 (102) | 0.609 (57.2)

17. Secondary Outcome: The Apparent Clearance of the Analyte in Plasma at Steady State Following Oral Administration (CL/F,ss) for PK Population (All Subjects)
Description: CL/F,ss = Apparent clearance of the analyte in the plasma at steady state following oral administration
Time Frame: 27 days
Population: PK Population - Subjects with values for CL/F,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 23 | 24 | 23 | 24
mL/min | 1007 (29.7) | 833 (21.5) | 1310 (113) | 1228 (104)

18. Secondary Outcome: The Apparent Clearance of the Analyte in Plasma at Steady State Following Oral Administration (CL/F,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: CL/F,ss = Apparent clearance of the analyte in the plasma at steady state following oral administration
Time Frame: 27 days
Population: PK Population excluding subjects with reported emesis - Subjects with values for CL/F,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 21 | 18 | 18
mL/min | 942 (19.6) | 839 (22.6) | 1008 (34.6) | 911 (40.4)

19. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase at Steady State Following Oral Administration (Vz/F,ss) for PK Population (All Subjects)
Description: Vz/F,ss = Apparent volume of distribution during the terminal phase λz at steady state following oral administration
Time Frame: 27 days
Population: PK Population - Subjects with values for Vz/F,ss
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 21 | 23 | 19 | 24
L | 1167 (50.3) | 545 (40.6) | 1671 (135) | 897 (138)

20. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase at Steady State Following Oral Administration (Vz/F,ss) for PK Population (Excluding Subjects Due to Emesis)
Description: Vz/F,ss = Apparent volume of distribution during the terminal phase λz at steady state following oral administration
Time Frame: 27 days
Population: PK Population excluding subjects with reported emesis - Subjects with values for Vz/F,ss excluding subjects with reported emesis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 0.375 mg q.d.ER | 0.125 mg t.i.d. IR | 1.5 mg q.d. ER | 0.5 mg t.i.d. IR
Number analyzed (Participants) | 19 | 20 | 14 | 18
L | 1092 (47.0) | 547 (43.2) | 1211 (37.8) | 625 (45.8)

ADVERSE EVENTS:
Time Frame: 27 days
Groups:
- 0.75 mg q.d. ER Up-titration; 0.75 mg q.d. ER Down-titration: 0.75mg once daily (q.d.) of oral extended release (ER) tablet of pramipexole
- 0.375 mg q.d.ER Down-titration: 0.375mg once daily (q.d.) of oral extended release (ER) tablet of pramipexole
Arm/Group | 0.375 mg q.d.ER | 0.75 mg q.d. ER Up-titration | 1.5 mg q.d. ER | 0.75 mg q.d. ER Down-titration | 0.375 mg q.d.ER Down-titration | 0.125 mg t.i.d. IR | 0.5 mg t.i.d. IR
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 14/24 | 9/24 | 12/24 | 6/24 | 0/24 | 8/24 | 14/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.375 mg q.d.ER (N=24) | 0.75 mg q.d. ER Up-titration (N=24) | 1.5 mg q.d. ER (N=24) | 0.75 mg q.d. ER Down-titration (N=24) | 0.375 mg q.d.ER Down-titration (N=24) | 0.125 mg t.i.d. IR (N=24) | 0.5 mg t.i.d. IR (N=24)
Dizziness (Nervous system disorders) | 4 | 3 | 3 | 0 | 0 | 0 | 5
Somnolence (Nervous system disorders) | 1 | 0 | 6 | 0 | 0 | 0 | 5
Headache (Nervous system disorders) | 0 | 4 | 2 | 0 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 3 | 5 | 0 | 0 | 1 | 6
Vomiting (Gastrointestinal disorders) | 4 | 1 | 4 | 0 | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0 | 1 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 5 | 0 | 2 | 2 | 0 | 5 | 2
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Electrocardiogram change (Investigations) | 1 | 1 | 0 | 3 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.